CLINICAL TRIAL: NCT04895280
Title: Effectiveness of Corticosteroid vs Ketorolac Shoulder Injections: a Prospective Double-Blinded Randomized Trial
Brief Title: Effectiveness of Corticosteroid vs Ketorolac Shoulder Injections
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of participants
Sponsor: Michael Khazzam (Other)
Responsible Party: Sponsor-Investigator, Michael Khazzam, ASSOC PROFESSOR -Orthopaedic Surgery, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU-2021-0232
Record Dates: First submitted 2021-05-12; First posted 2021-05-20 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Full-thickness Rotator Cuff Tear; Rotator Cuff Tendinitis
Keywords: Shoulder; Rotator Cuff
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Ketorolac; Ketorolac Tromethamine; Bupivacaine; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (marcaine) (Other): will receive an injection of 4 cc 0.25% Marcaine without epinephrine
  Interventions: Drug: Marcaine
- Group 2 (ketorolac) (Experimental): will receive an injection of 4 cc 0.25% Marcaine without epinephrine and 30 mg ketorolac x 1
  Interventions: Drug: Ketorolac; Drug: Marcaine
- Group 3 (kenalog) (Other): 4 cc 0.25% Marcaine without epinephrine and 40 mg triamcinolone x 1. Group 3 is standard of care
  Interventions: Drug: Marcaine; Drug: Kenalog

INTERVENTIONS:
Drug: Ketorolac — Ketorolac: will receive an injection of 4 cc 0.25% Marcaine without epinephrine and 30 mg ketorolac x 1
  Other Names: Toradol
  Arms: Group 2 (ketorolac)
Drug: Marcaine — Marcaine (control): will receive an injection of 4 cc 0.25% Marcaine without epinephrine
  Other Names: Bupivacaine Hydrochloride
Drug: Kenalog — Kenalog: 4 cc 0.25% Marcaine without epinephrine and 40 mg triamcinolone x 1.
  Other Names: Triamcinolone Acetonide
  Arms: Group 3 (kenalog)

SUMMARY:
The purpose of this study is to compare the functional outcomes of patients with shoulder pathology treated with either ketorolac or corticosteroid injections, in a randomized double-blinded study. Investigators will compare the effectiveness of ketorolac compared to corticosteroid.

Specific Aim 1:

Hypothesis 1: Injection of the shoulder (in the subacromial space) with Ketorolac will be more effective than corticosteroid injection for the treatment of a variety of shoulder pathologies.

The risks associated with this study primarily concern adverse reactions to the study drugs. The drugs used in this study are not narcotics or habit-forming but can have side effects. The patient's physician will screen for any heart, intestinal, or kidney disease or condition that would increase the chance for the patient to have an unwanted side effect.

DETAILED DESCRIPTION:
The proposed study is a three arm, double-blinded, prospective randomized controlled clinical trial with follow-up immediately after the injection and at day 2, and weeks 1, 2, 4, 6, and 12. In this study investigators will compare the effectiveness of ketorolac compared to corticosteroid.

Subjects being seen for a rotator cuff injury will be randomized into one of three treatment groups pertaining to their pathology. The intervention will begin once the subject has consented and answered the Baseline Outcome Shoulder Questionnaire. The Baseline Outcome Questionnaire consists of the Visual Analog Score, American Shoulder and Elbow Score, Single Assessment Numeric Evaluation, Pittsburgh Sleep Quality Index, Short Form-12, and questions pertaining to patient characteristics, injury characteristics, co-morbidities, patient history, medications, and demographics.

ELIGIBILITY:
Inclusion Criteria:

* Age: > or = 18 years old
* Rotator Cuff Tendinitis
* Atraumatic Full-thickness Rotator Cuff Tear
* Subjects who speak English
* Women who are of non-childbearing potential

Exclusion Criteria:

* Age: < 18 years old
* Prior Shoulder Surgery
* Fracture
* Acute Traumatic Rotator Cuff Tear
* Infection
* Uncontrolled Diabetes Mellitus (HbA1c >8)
* Uncontrolled High Blood Pressure (Hypertension)
* Recent Prior Shoulder Injection in either the Subacromial space Workers Compensation
* History of Peptic Ulcer disease (includes both Gastric and Duodenal Ulcers), Gastrointestinal perforation, Inflammatory Bowel disease (Ulcerative Colitis, Crohn's disease), or any other gastrointestinal pathology
* Tumor Involving the Shoulder Region
* Prior history of gastrointestinal bleeding, allergic reactions, impaired renal function, seizures or cardiac arrhythmias
* Subject unable to provide informed consent
* Subjects who don't speak English
* Patients who are pregnant or lactating at time of screening or are of pregnant bearing age
* Patients currently receiving an aspirin, NSAID regimen or any other anti-inflammatory agents that could affect inflammation response.
* Patients taking any anti-platelet agents, warfarin or other anticoagulants, or SSRIs.
* Patients with any bleeding disorders such as coagulopathy, hypercoagulable state, or platelet disorders including thrombocytopenia.
* Patients with cardiac disease such as congestive heart failure, coronary artery disease, or myocardial infarction.
* Patients with severe renal failure. Patients with severe liver impairment or active liver disease.
* Patients with heavy alcohol use; this is defined as consuming 8 or more drinks per week for a woman and 15 or more drinks per week for a man.
* Patients likely to have severe problems maintaining follow-up, including patients diagnosed with severe psychiatric conditions, patients who live too far outside the hospital's catchment area, patients who are incarcerated and patients who have unstable housing situations. Patients with a known hypersensitivity to bupivacaine or other local anesthetic agent of the amide-type.
* Patients who have experienced asthma, urticaria, or allergic-type reactions after taking aspirin or other NSAIDs
* Patients who are allergic to aspirin, ketorolac tromethamine and other NSAIDs.
* Patients who are currently on probenecid or pentoxifylline as described in the approved label of Ketorolac tromethamine injection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | Baseline - pre-injection
  Pain as measured by the Visual Analog Scale prior to first injection. The visual analog scale is a 0-10 scale, 0 being no pain, 10 being unbearable pain.
Visual Analog Scale | Baseline - immediately after the injection
  Pain as measured by the Visual Analog Scale after first injection. The visual analog scale is a 0-10 scale, 0 being no pain, 10 being unbearable pain.
Visual Analog Scale | Day 2
  Pain as measured by the Visual Analog Scale. The visual analog scale is a 0-10 scale, 0 being no pain, 10 being unbearable pain.
Visual Analog Scale | Week 1
  Pain as measured by the Visual Analog Scale. The visual analog scale is a 0-10 scale, 0 being no pain, 10 being unbearable pain.
Visual Analog Scale | Week 2
  Pain as measured by the Visual Analog Scale. The visual analog scale is a 0-10 scale, 0 being no pain, 10 being unbearable pain.
Visual Analog Scale | Week 4
  Pain as measured by the Visual Analog Scale. The visual analog scale is a 0-10 scale, 0 being no pain, 10 being unbearable pain.
Visual Analog Scale | Week 6
  Pain as measured by the Visual Analog Scale. The visual analog scale is a 0-10 scale, 0 being no pain, 10 being unbearable pain.
Visual Analog Scale | Week 12
  Pain as measured by the Visual Analog Scale. The visual analog scale is a 0-10 scale, 0 being no pain, 10 being unbearable pain.
American Shoulder and Elbow Score (ASES) | Baseline
  Pain, instability, and activities of daily living as measured by the American Shoulder and Elbow Score. The ASES is a 100-point scale that consists of two dimensions: pain and activities of daily living. One pain scale is worth 50 points, and activities of daily living worth 50 points. A higher score indicates a better outcome.
American Shoulder and Elbow Score (ASES) | Week 6
  Pain, instability, and activities of daily living as measured by the American Shoulder and Elbow Score. The ASES is a 100-point scale that consists of two dimensions: pain and activities of daily living. One pain scale is worth 50 points, and activities of daily living worth 50 points. A higher score indicates a better outcome.
American Shoulder and Elbow Score (ASES) | Week 12
  Pain, instability, and activities of daily living as measured by the American Shoulder and Elbow Score. The ASES is a 100-point scale that consists of two dimensions: pain and activities of daily living. One pain scale is worth 50 points, and activities of daily living worth 50 points. A higher score indicates a better outcome.

SECONDARY OUTCOMES:
Single Assessment Numeric Evaluation (SANE) | Baseline
  Measure the patient's self-reported function on a scale of 0 to 100
Single Assessment Numeric Evaluation (SANE) | Week 6
  Measure the patient's self-reported function on a scale of 0 to 100
Single Assessment Numeric Evaluation (SANE) | Week 12
  Measure the patient's self-reported function on a scale of 0 to 100
Pittsburgh Sleep Quality Index (PSQI) | Baseline
  Sleep quality as measured by the Pittsburgh Sleep Quality Index
Pittsburgh Sleep Quality Index (PSQI) | Week 6
  Sleep quality as measured by the Pittsburgh Sleep Quality Index
Pittsburgh Sleep Quality Index (PSQI) | Week 12
  Sleep quality as measured by the Pittsburgh Sleep Quality Index
Short Form 12 (SF-12) | Baseline
  General health survey as measured by the Short Form 12 (SF-12)
Short Form 12 (SF-12) | Week 6
  General health survey as measured by the Short Form 12 (SF-12)
Short Form 12 (SF-12) | Week 12
  General health survey as measured by the Short Form 12 (SF-12)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Khazzam, MD, Principal Investigator — 214-645-3300
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adebajo AO, Nash P, Hazleman BL. A prospective double blind dummy placebo controlled study comparing triamcinolone hexacetonide injection with oral diclofenac 50 mg TDS in patients with rotator cuff tendinitis. J Rheumatol. 1990 Sep;17(9):1207-10. PMID 2290163
- [Background] Alvarez CM, Litchfield R, Jackowski D, Griffin S, Kirkley A. A prospective, double-blind, randomized clinical trial comparing subacromial injection of betamethasone and xylocaine to xylocaine alone in chronic rotator cuff tendinosis. Am J Sports Med. 2005 Feb;33(2):255-62. doi: 10.1177/0363546504267345. PMID 15701612
- [Background] Choi WD, Cho DH, Hong YH, Noh JH, Lee ZI, Byun SD. Effects of subacromial bursa injection with corticosteroid and hyaluronidase according to dosage. Ann Rehabil Med. 2013 Oct;37(5):668-74. doi: 10.5535/arm.2013.37.5.668. Epub 2013 Oct 29. PMID 24236254
- [Background] Blair B, Rokito AS, Cuomo F, Jarolem K, Zuckerman JD. Efficacy of injections of corticosteroids for subacromial impingement syndrome. J Bone Joint Surg Am. 1996 Nov;78(11):1685-9. doi: 10.2106/00004623-199611000-00007. PMID 8934482
- [Background] Min KS, St Pierre P, Ryan PM, Marchant BG, Wilson CJ, Arrington ED. A double-blind randomized controlled trial comparing the effects of subacromial injection with corticosteroid versus NSAID in patients with shoulder impingement syndrome. J Shoulder Elbow Surg. 2013 May;22(5):595-601. doi: 10.1016/j.jse.2012.08.026. Epub 2012 Nov 22. PMID 23177167
- [Background] Penning LI, de Bie RA, Walenkamp GH. The effectiveness of injections of hyaluronic acid or corticosteroid in patients with subacromial impingement: a three-arm randomised controlled trial. J Bone Joint Surg Br. 2012 Sep;94(9):1246-52. doi: 10.1302/0301-620X.94B9.28750. PMID 22933498
- [Background] Karthikeyan S, Kwong HT, Upadhyay PK, Parsons N, Drew SJ, Griffin D. A double-blind randomised controlled study comparing subacromial injection of tenoxicam or methylprednisolone in patients with subacromial impingement. J Bone Joint Surg Br. 2010 Jan;92(1):77-82. doi: 10.1302/0301-620X.92B1.22137. PMID 20044683
- [Background] Koester MC, Dunn WR, Kuhn JE, Spindler KP. The efficacy of subacromial corticosteroid injection in the treatment of rotator cuff disease: A systematic review. J Am Acad Orthop Surg. 2007 Jan;15(1):3-11. doi: 10.5435/00124635-200701000-00002. PMID 17213378
- [Background] Marder RA, Kim SH, Labson JD, Hunter JC. Injection of the subacromial bursa in patients with rotator cuff syndrome: a prospective, randomized study comparing the effectiveness of different routes. J Bone Joint Surg Am. 2012 Aug 15;94(16):1442-7. doi: 10.2106/JBJS.K.00534. PMID 22992814
- [Background] Balasubramaniam P, Prathap K. The effect of injection of hydrocortisone into rabbit calcaneal tendons. J Bone Joint Surg Br. 1972 Nov;54(4):729-34. No abstract available. PMID 4639447
- [Background] Kapetanos G. The effect of the local corticosteroids on the healing and biomechanical properties of the partially injured tendon. Clin Orthop Relat Res. 1982 Mar;(163):170-9. PMID 7067249
- [Background] Oxlund H. The influence of a local injection of cortisol on the mechanical properties of tendons and ligaments and the indirect effect on skin. Acta Orthop Scand. 1980 Apr;51(2):231-8. doi: 10.3109/17453678008990791. PMID 7435179
- [Background] Wiggins ME, Fadale PD, Barrach H, Ehrlich MG, Walsh WR. Healing characteristics of a type I collagenous structure treated with corticosteroids. Am J Sports Med. 1994 Mar-Apr;22(2):279-88. doi: 10.1177/036354659402200221. PMID 8198200
- [Background] Wei AS, Callaci JJ, Juknelis D, Marra G, Tonino P, Freedman KB, Wezeman FH. The effect of corticosteroid on collagen expression in injured rotator cuff tendon. J Bone Joint Surg Am. 2006 Jun;88(6):1331-8. doi: 10.2106/JBJS.E.00806. PMID 16757768
- [Background] Dogan N, Erdem AF, Gundogdu C, Kursad H, Kizilkaya M. The effects of ketorolac and morphine on articular cartilage and synovium in the rabbit knee joint. Can J Physiol Pharmacol. 2004 Jul;82(7):502-5. doi: 10.1139/y04-066. PMID 15389297
- [Background] Jean YH, Wen ZH, Chang YC, Hsieh SP, Tang CC, Wang YH, Wong CS. Intra-articular injection of the cyclooxygenase-2 inhibitor parecoxib attenuates osteoarthritis progression in anterior cruciate ligament-transected knee in rats: role of excitatory amino acids. Osteoarthritis Cartilage. 2007 Jun;15(6):638-45. doi: 10.1016/j.joca.2006.11.008. Epub 2007 Jan 2. PMID 17198754
- [Background] Itzkowitch D, Ginsberg F, Leon M, Bernard V, Appelboom T. Peri-articular injection of tenoxicam for painful shoulders: a double-blind, placebo controlled trial. Clin Rheumatol. 1996 Nov;15(6):604-9. doi: 10.1007/BF02238552. PMID 8973872
- [Background] Kenaolg Package Insert. July 2014; Available from: http://packageinserts.bms.com/pi/pi_kenalog-40.pdf.
- [Background] Ketorolac: Drug Class and Mechanism. 2014; Available from: http://www.medicinenet.com/ketorolac-oral/article.htm
- [Background] Ogbru, O. Marcaine - Drug Class and Mechanism. 6/27/2014; Available from: http://www.medicinenet.com/bupivicaine-injection/article.htm.
- [Background] Kenalog: Drug Summary. Available from: http://www.pdr.net/drug-summary/kenalog-40?druglabelid=2494
- [Background] Hawker, G.A., et al. Measures of Adult Pain. 2011; Available from: http://onlinelibrary.wiley.com/doi/10.1002/acr.20543/pdf
- [Background] Gould D, Kelly D, Goldstone L, Gammon J. Examining the validity of pressure ulcer risk assessment scales: developing and using illustrated patient simulations to collect the data. J Clin Nurs. 2001 Sep;10(5):697-706. doi: 10.1046/j.1365-2702.2001.00525.x. PMID 11822520
- [Background] Michener LA, McClure PW, Sennett BJ. American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form, patient self-report section: reliability, validity, and responsiveness. J Shoulder Elbow Surg. 2002 Nov-Dec;11(6):587-94. doi: 10.1067/mse.2002.127096. PMID 12469084
- [Background] Richards RR, An KN, Bigliani LU, Friedman RJ, Gartsman GM, Gristina AG, Iannotti JP, Mow VC, Sidles JA, Zuckerman JD. A standardized method for the assessment of shoulder function. J Shoulder Elbow Surg. 1994 Nov;3(6):347-52. doi: 10.1016/S1058-2746(09)80019-0. Epub 2009 Feb 13. PMID 22958838
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Gerstenfeld LC, Al-Ghawas M, Alkhiary YM, Cullinane DM, Krall EA, Fitch JL, Webb EG, Thiede MA, Einhorn TA. Selective and nonselective cyclooxygenase-2 inhibitors and experimental fracture-healing. Reversibility of effects after short-term treatment. J Bone Joint Surg Am. 2007 Jan;89(1):114-25. doi: 10.2106/JBJS.F.00495. PMID 17200318
- [Background] Ho ML, Chang JK, Wang GJ. Effects of ketorolac on bone repair: A radiographic study in modeled demineralized bone matrix grafted rabbits. Pharmacology. 1998 Sep;57(3):148-59. doi: 10.1159/000028236. PMID 9691235
- [Background] O'Keefe RJ, Tiyapatanaputi P, Xie C, Li TF, Clark C, Zuscik MJ, Chen D, Drissi H, Schwarz E, Zhang X. COX-2 has a critical role during incorporation of structural bone allografts. Ann N Y Acad Sci. 2006 Apr;1068:532-42. doi: 10.1196/annals.1346.012. PMID 16831949
- [Background] Haws MJ, Kucan JO, Roth AC, Suchy H, Brown RE. The effects of chronic ketorolac tromethamine (toradol) on wound healing. Ann Plast Surg. 1996 Aug;37(2):147-51. doi: 10.1097/00000637-199608000-00005. PMID 8863973
- [Background] Prisk V, Huard J. Muscle injuries and repair: the role of prostaglandins and inflammation. Histol Histopathol. 2003 Oct;18(4):1243-56. doi: 10.14670/HH-18.1243. PMID 12973691
- [Background] Radi ZA, Khan NK. Effects of cyclooxygenase inhibition on bone, tendon, and ligament healing. Inflamm Res. 2005 Sep;54(9):358-66. doi: 10.1007/s00011-005-1367-4. PMID 16273333
- [Background] Sucato DJ, Lovejoy JF, Agrawal S, Elerson E, Nelson T, McClung A. Postoperative ketorolac does not predispose to pseudoarthrosis following posterior spinal fusion and instrumentation for adolescent idiopathic scoliosis. Spine (Phila Pa 1976). 2008 May 1;33(10):1119-24. doi: 10.1097/BRS.0b013e31816f6a2a. PMID 18449047
- [Background] Pradhan BB, Tatsumi RL, Gallina J, Kuhns CA, Wang JC, Dawson EG. Ketorolac and spinal fusion: does the perioperative use of ketorolac really inhibit spinal fusion? Spine (Phila Pa 1976). 2008 Sep 1;33(19):2079-82. doi: 10.1097/BRS.0b013e31818396f4. PMID 18698276
- [Background] Glassman SD, Rose SM, Dimar JR, Puno RM, Campbell MJ, Johnson JR. The effect of postoperative nonsteroidal anti-inflammatory drug administration on spinal fusion. Spine (Phila Pa 1976). 1998 Apr 1;23(7):834-8. doi: 10.1097/00007632-199804010-00020. PMID 9563116
- [Background] Park SY, Moon SH, Park MS, Oh KS, Lee HM. The effects of ketorolac injected via patient controlled analgesia postoperatively on spinal fusion. Yonsei Med J. 2005 Apr 30;46(2):245-51. doi: 10.3349/ymj.2005.46.2.245. PMID 15861498
- [Background] Mullis BH, Copland ST, Weinhold PS, Miclau T, Lester GE, Bos GD. Effect of COX-2 inhibitors and non-steroidal anti-inflammatory drugs on a mouse fracture model. Injury. 2006 Sep;37(9):827-37. doi: 10.1016/j.injury.2005.12.018. Epub 2006 Feb 23. PMID 16497308